CLINICAL TRIAL: NCT01221831
Title: A Randomised Open-label Multi-centre Comparative Study to Evaluate Cycle Control of 2 Dosages of Estetrol Combined With Either P1 or P2, Compared to a Combined Oral Contraceptive Containing E2V and DNG
Brief Title: Cycle Control Assessment of a Combined Oral Contraceptive Containing Estetrol and a Progestin P1 or P2
Acronym: FIESTA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Estetra (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ES-C02; 2010-019865-26 (EudraCT Number)
Record Dates: First submitted 2010-10-13; First posted 2010-10-15 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Contraception
MeSH Terms: interventions — Estetrol; P-2; Estradiol; dienogest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- estetrol dose 1 / P1 (Experimental)
  Interventions: Drug: estetrol, P 1 and placebo tablets
- estetrol dose 1 / P2 (Experimental)
  Interventions: Drug: estetrol, P2 and placebo tablets
- estradiol valerate/dienogest pill (Active Comparator)
  Interventions: Drug: Estradiol valerate, dienogest and placebo tablets
- estetrol dose 2 / P1 (Experimental)
  Interventions: Drug: estetrol, P 1 and placebo tablets
- estetrol dose 2 / P2 (Experimental)
  Interventions: Drug: estetrol, P2 and placebo tablets

INTERVENTIONS:
Drug: estetrol, P 1 and placebo tablets — 6 treatment cycles each consisting of 28 days of oral administration as follows:
  * Days 1-24: one estetrol tablet and one P1 tablet per day
  * Days 25-28: two placebo tablets per day
  Arms: estetrol dose 1 / P1; estetrol dose 2 / P1
Drug: estetrol, P2 and placebo tablets — 6 treatment cycles each consisting of 28 days of oral administration as follows:
  * Days 1-24: one estetrol tablet and one P2 tablet per day
  * Days 25-28: two placebo tablets per day
  Arms: estetrol dose 1 / P2; estetrol dose 2 / P2
Drug: Estradiol valerate, dienogest and placebo tablets — 6 treatment cycles each consisting of 28 days of oral administration as follows:
  * Days 1-26: one tablet of Estradiol valerate/dienogest per day
  * Days 26-28: one placebo tablet per day
  Arms: estradiol valerate/dienogest pill

SUMMARY:
This is an open-label, multi-centre, comparative study in young, healthy, female volunteers of reproductive age.

Primary objective:

- To investigate the effect of 2 dosages of estetrol combined with P1 or P2, on vaginal bleeding patterns (cycle control), in comparison with a combined oral contraceptive containing estradiol valerate and dienogest

Secondary objectives:

* To investigate ovulation inhibition
* To investigate the effect on SHBG
* To assess pregnancy rate
* To evaluate subject satisfaction, dysmenorrhoea, acne, and body weight
* To investigate return of menstruation after treatment
* To evaluate general safety and acceptability

ELIGIBILITY:
Inclusion Criteria:

* Women willing to use a Combined Oral Contraceptive for 6 subsequent cycles
* Good physical and mental health
* Regular menstrual cycle (24-35 days) prior to screening
* Body mass index between (≥) 18 and (≤) 30 kg/m2

Exclusion Criteria:

* Previous use of any hormonal contraceptive method during the last 3 months prior to randomisation (only applicable for women who are not using a hormonal contraceptive method at the time of screening)
* Previous use of progestogen-only contraceptive methods during the last 3 months or during the last 6 months for depot progestogen preparations or an injectable hormonal method of contraception
* Use of phytoestrogens
* No spontaneous menstruation has occurred following a delivery or abortion
* Breastfeeding or within 2 months after stopping breastfeeding prior to the start of study medication and no spontaneous return of menstruation
* Status post-partum or post-abortion within a period of 2 months before screening
* Pregnancy during accurate hormonal contraceptive use in the past
* Intention to become pregnant during the study
* An abnormal cervical smear within one year before study start
* Untreated Chlamydia infection
* Known or suspected breast cancer or a history of breast cancer
* A history of (within 12 months) alcohol or drug abuse
* Any clinically relevant abnormality
* Contraindications for the contraceptive steroids used in the clinical trial
* Use of antihypertensive drugs or use of medications interacting with the contraceptive steroids used in the clinical trial
* Administration of any other investigational drug within 2 months prior to screening

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 396 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Recording of vaginal bleeding events (diary) as a measure of Cycle control | 6 cycles of 28 days

SECONDARY OUTCOMES:
Measurement of pregnandiol glucuronide in urine as a measure of Ovulation inhibition | 6 cycles of 28 days
Patient Reported Outcome questionnaire as a measure of Subject satisfaction | 6 cycles of 28 days
Contacts patient-investigator to document Return of menstruation | for up to 1 year follow-up
  (only in case the patient does not start up a new hormonal contraceptive method or in case of pregnancy wish)
Recording of adverse events, physical examination and laboratory parameters as a measure of Safety and Tolerability | up to 8 months
Measurement of SHBG in blood samples to assess the effect of treatment on SHBG | 6 cycles of 28 days
Reporting of in-treatment pregnancies as a measure of pregnancy rate | 6 cycles of 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Dan Apter, M.D., Principal Investigator — Väestöliitto Helsinki
Locations (10):
- Finland (10):
  - Mehiläinen Helsinki, Helsinki
  - Väestöliitto Helsinki, Helsinki
  - YTHS Jyvaskyla, Jyväskylä
  - Laboratorio Simpanen, Kuopio
  - Terveystalo Kuopio, Kuopio
  - YTHS Kuopio, Kuopio
  - Väestöliitto Oulu, Oulu
  - Tampereen Lääkärikeskus Oy, Tampere
  - YTHS Tampere, Tampere
  - Väestöliitto Turku, Turku